CLINICAL TRIAL: NCT00022074
Title: Control of Vasomotor Symptoms in Women Treated for Breast Cancer
Brief Title: Gabapentin For the Control of Hot Flashes in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Morrow, Director, University of Rochester NCORP Research Base, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000068780; URCC-U2101; NCI-P01-0183
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Anxiety Disorder; Breast Cancer; Depression; Hot Flashes
Keywords: stage I breast cancer; stage II breast cancer; stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; anxiety disorder; depression; hot flashes
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms; Depression; Hot Flashes | interventions — Gabapentin

INTERVENTIONS:
Drug: gabapentin
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Gabapentin may be effective for the control of hot flashes. It is not yet known if gabapentin is effective in treating hot flashes.

PURPOSE: Randomized clinical trial to study the effectiveness of gabapentin in controlling hot flashes in women who have breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effectiveness and side effects of 2 different doses of gabapentin vs placebo for the control of hot flashes and other vasomotor symptoms in women with breast cancer.
* Compare quality of life, anxiety, and depression in patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to participating center and duration of hot flash symptoms (less than 9 months vs 9 or more months). Patients are randomized to 1 of 3 arms.

* Arm I: Patients receive oral placebo 3 times a day.
* Arm II: Patients receive oral gabapentin at a low dose 3 times a day.
* Arm III: Patients receive oral gabapentin as in arm II for 3 days and then at a high dose 3 times a day.

Treatment on all arms continues for 8 weeks in the absence of unacceptable toxicity. After week 8, patients may receive open-label gabapentin at the discretion of their physicians.

Hot flashes are assessed at baseline and then during weeks 3 and 7 of the study.

Quality of life, anxiety, and depression are assessed at baseline and then at weeks 4 and 8.

Patients are followed at week 12.

PROJECTED ACCRUAL: A total of 408 patients (136 per arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer
* Experiencing 2 or more hot flashes per day for at least 1 week
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Not specified

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin normal
* SGOT no greater than 2 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 1.25 times ULN

Cardiovascular:

* No coronary insufficiency
* No myocardial infarction within the past 3 months
* No symptomatic cardiac disease
* No peripheral vascular disease
* No cerebrovascular disease or stroke
* No syncope or symptomatic hypotension

Other:

* No history of allergic or other adverse reaction to gabapentin
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 1 week after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No other concurrent anticonvulsant medication
* No concurrent clonidine or venlafaxine

Max Age: 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-07; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kishan J. Pandya, MD, Study Chair — James P. Wilmot Cancer Center
Locations (18):
- United States (18):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - CCOP - North Shore University Hospital, Manhasset, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin

REFERENCES:
- [Result] Pandya KJ, Morrow GR, Roscoe JA, Zhao H, Hickok JT, Pajon E, Sweeney TJ, Banerjee TK, Flynn PJ. Gabapentin for hot flashes in 420 women with breast cancer: a randomised double-blind placebo-controlled trial. Lancet. 2005 Sep 3-9;366(9488):818-24. doi: 10.1016/S0140-6736(05)67215-7. PMID 16139656